CLINICAL TRIAL: NCT00908375
Title: Efficacy of Pregabalin in Patients With Radicular Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, kahlid malik, Assistant Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRA7057
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2014-09-16 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-09

CONDITIONS: Neuropathy; Radicular, Lumbar, Lumbosacral; Failed Back Surgery Syndrome; Spinal Stenosis; Herniated Disc
Keywords: Pregabalin; Radicular pain; Failed back surgery; Of greater than 3 months duration
MeSH Terms: conditions — Failed Back Surgery Syndrome; Spinal Stenosis; Intervertebral Disc Displacement | interventions — Pregabalin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Active Comparator): A 75mg pregabalin capsule will be prescribed twice daily for the first week of the study (150mg/day). For the subsequent 2 weeks, the dose will be increased to 2 pregabalin capsules twice a day (300mg/day). The total duration of the treatment will be 3 weeks.
  Interventions: Drug: Pregabalin
- Surgar Pill (Placebo Comparator): One Sugar pill capsule will be prescribed twice daily for the first week of the study. For the subsequent 2 weeks, 2 Sugar pill capsules twice a day. The total duration of the treatment will be 3 weeks.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Pregabalin — One pregabalin 75mg capsule will be prescribed twice daily for the first week of the study (150mg/day). For the subsequent 2 weeks, the dose will be increased to 2 pregabalin capsules twice a day (300mg/day). The total duration of the treatment will be 3 weeks.
  Other Names: Lyrica®, Pfizer NY, NY 10017
  Arms: Pregabalin
Drug: Sugar Pill — One sugar pill will be prescribed twice daily for the first week of the study. For the subsequent 2 weeks, 2 placebo(sugar pills) capsules twice a day. The total duration of the treatment will be 3 weeks.
  Other Names: Placebo
  Arms: Surgar Pill

SUMMARY:
The purpose of this study is to evaluate whether pregabalin is effective in reducing the pain in patients who present with radicular pain due to a herniated disc, spinal stenosis or failed back surgery syndrome.

DETAILED DESCRIPTION:
Although the efficacy of pregabalin has been demonstrated in several pain states and it is approved by the FDA for use in post herpetic neuralgia, diabetic neuropathy and fibromyalgia there are few studies of its efficacy in patients with radicular pain from herniated disc, spinal stenosis or failed back surgery syndrome. This study was conducted to evaluate the efficacy of pregabalin in these pain states.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pain in dermatomal distribution, in either cervical or lumbar region.
2. History of pain for more than 3 months.
3. History of herniated disc, spinal stenosis or failed back surgery.
4. A series of epidural steroid injections within the past 6 months.
5. Presence of motor or sensory neurological signs (hypoesthesia, hyperesthesia, allodynia, dysesthesia) in the affected dermatomes.
6. Patients must be cognitively capable of completing the pain questionnaires.

Exclusion Criteria:

1. Patients below 18 or over 65 years of age.
2. Patients with mostly axial spinal pain.
3. Presence of significant motor deficits, and /or bowel and/or bladder dysfunction.
4. Workmen's compensation or disability issues.
5. Patients with chronic depression and on depression medications.
6. Addiction and/or substance abuse issues.
7. Patients using gabapentin or failure to respond to previous gabapentin use.
8. Patients with known peripheral neuropathy (e.g. DPN, PHN etc.).
9. Known hypersensitivity to pregabalin use (hives, blisters, rash, dypnea and wheezing).
10. History of angioedema with pregabalin use.
11. Patients with known renal insufficiency, diabetes, congestive heart failure, cardiac conduction abnormalities, and/or thrombocytopenia.
12. Patients using ACE-inhibitors and thiazolidinedione antidiabetic agents (Avandia®, Actos®).
13. Pregnant patients.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khalid M Malik, MD, Principal Investigator — Northwestern University
Locations (1):
- Pain Medicine Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: One Sugar pill capsule will be prescribed twice daily for the first week of the study. For the subsequent 2 weeks, 2 Sugar pill capsules twice a day. The total duration of the treatment will be 3 weeks.
  Sugar Pill: One sugar pill will be prescribed twice daily for the first week of the study. For the subsequent 2 weeks, 2 placebo(sugar pills) capsules twice a day. The total duration of the treatment will be 3 weeks.
Period: Overall Study
Arm/Group | Pregabalin | Sugar Pill
Started | 20 | 19
Completed | 10 | 9
Not Completed | 10 | 10
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Sugar Pill | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10.17) | 44 (13.38) | 45 (11.78)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 9 | 11 | 20
Pain Score (Numeric Rating Scale , 0-10) [Median (Inter-Quartile Range); unit: units on a scale] — Numeric Rating Pain scale ranging from 0 (no pain) to 10 (worst pain imaginable).
  units on a scale | 6.5 [4.5 to 7] | 6 [3 to 7] | 6 [4 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores (NRS) at 3-weeks
Description: Standard numeric rating pain scale ranging from 0 (no pain) to 10 (worst pain imaginable) after 3 weeks of treatment.
  .
Time Frame: 3 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pregabalin | Sugar Pill
Number analyzed (Participants) | 10 | 9
units on a scale | 6 [1 to 9] | 3 [0 to 8]
Statistical Analysis 1: Comparison: Pregabalin vs Sugar Pill; Test type: Non-Inferiority or Equivalence — Sample size was determined based on the primary outcome variable, the VAS pain score at three weeks. Based on the results of the study of Siddall et al., group sample sizes of 19 and 19 achieve 82% power to detect a difference of 2.00 between the null hypothesis that both group means are 6.50 and the alternative hypothesis that the mean of pregabalin group is 4.50 with estimated group standard deviations of 2.10 and 2.10 and with a significance level of 0.05 using a two-sided two-sample t-test; p = 0.279, Wilcoxon (Mann-Whitney) — The criterion for rejection of the null hypothesis (P < 0.05) was adjusted for multiple application of the test to the same data set using the Bonferroni correction; Median Difference (Final Values) = -2, 99% CI 2-sided [-6 to 3]

2. Secondary Outcome: Patient's Global Impression of Change at 3 Weeks
Description: Global impression of change in patient status reported at 3 weeks. The global impression of change consists of a Likert scale as below:
  1. Very Much Improved
  2. Much Improved
  3. Minimally Improved
  4. No Change
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
Time Frame: 3 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pregabalin | Sugar Pill
Number analyzed (Participants) | 10 | 9
units on a scale | 3.5 [1 to 5] | 3 [1 to 4]
Statistical Analysis 1: Comparison: Pregabalin vs Sugar Pill; Test type: Superiority or Other; p = 0.282, Wilcoxon (Mann-Whitney) — The criterion for rejection of the null hypothesis (P < 0.05) was adjusted for multiple applications of the test to the same data using the Bonferroni correction; Median Difference (Final Values) = -1, 99% CI 2-sided [-2.0 to 1.0]

3. Secondary Outcome: Oswestry Disability Questionnaires
Description: Oswestry disability index (ODI) is a tool to measure a subject's functional disability. The Oswestry disability index consists of 10 questions with a Likert 0-5 scale. Each individual score is converted into a percent which represents the "percent disability." There are five tiers, 0-20% (minimal disability), 21%-40% (moderate disability), 41%-60% (severe disability), 61%-80% (crippled), 81%-100% (i.e. bed bound). We report the Oswestry disability scores at 3 weeks.
Time Frame: 3 weeks
Measure: Median (Full Range); unit: percent disability
Arm/Group | Pregabalin | Sugar Pill
Number analyzed (Participants) | 10 | 9
percent disability | 41 [8 to 64] | 20 [2 to 60]
Statistical Analysis 1: Comparison: Pregabalin vs Sugar Pill; Test type: Superiority or Other; p = 0.139, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -16, 99% CI 2-sided [-42 to 16]

ADVERSE EVENTS:
Time Frame: Subject reported difficulty in swallowing sensation 4 days following the start of the study. Symptoms resolved within 48 hrs following discontinuation of the study drug.
Arm/Group | Pregabalin | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=20) | Sugar Pill (N=19)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Exacerbation of existing migraine headache

LIMITATIONS AND CAVEATS:
Early subject withdrawal and lost to follow-up leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes